CLINICAL TRIAL: NCT07113145
Title: Comparative Evaluation of Safety and Efficacy of Dapoxetine, Silodosin, and Citalopram in the Management of Premature Ejaculation: A Randomized Clinical Trial
Brief Title: Comparative Evaluation of Safety and Efficacy of Dapoxetine, Silodosin, and Citalopram in the Management of Premature Ejaculation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdallah, lecturer of urology, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMBSUREC/07052024/Ahmed
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Premature (Early) Ejaculation
Keywords: Premature ejaculation; Citalopram; Dapoxetine; Silodosin; IELT; PEPQ
MeSH Terms: conditions — Premature Birth; Premature Ejaculation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Received Citalopram, starting with 10 mg once daily for 1 week, followed by 20 for 10 weeks (Active Comparator)
  Interventions: Drug: Oral intake of medication
- Received Silodosin 4mg, administered orally once daily. (Active Comparator)
  Interventions: Drug: Oral intake of medication
- Received Dapoxetine 30 mg, taken 2 hours before intercourse, on-demand, min 8/ month for 3 mon (Active Comparator)
  Interventions: Drug: Oral intake of medication
- Received Dapoxetine hydrochloride 30 mg, administered daily. (Active Comparator)
  Interventions: Drug: Oral intake of medication

INTERVENTIONS:
Drug: Oral intake of medication — ● Group A: Received Citalopram hydrobromide, starting with 10 mg once daily for 1 week, followed by 20 mg once daily for 10 weeks, and 10 mg daily during the final week (tapered).
  Arms: Received Citalopram, starting with 10 mg once daily for 1 week, followed by 20 for 10 weeks
Drug: Oral intake of medication — ● Group B: Received Silodosin 4mg, administered orally once daily.
  Arms: Received Silodosin 4mg, administered orally once daily.
Drug: Oral intake of medication — ● Group C: Received Dapoxetine hydrochloride 30 mg, taken 2 hours before intercourse, on-demand, minimum of 8 times/month for 3 months.
  Arms: Received Dapoxetine 30 mg, taken 2 hours before intercourse, on-demand, min 8/ month for 3 mon
Drug: Oral intake of medication — ● Group D: Received Dapoxetine hydrochloride 30 mg, administered daily.
  Arms: Received Dapoxetine hydrochloride 30 mg, administered daily.

SUMMARY:
This randomized controlled trial evaluated the comparative effectiveness and safety of four pharmacological treatments-Citalopram 20mg, Silodosin 4 mg, Dapoxetine 30 mg on demand, and Dapoxetine 30 mg daily-in men with premature ejaculation (PE). A total of 400 male patients were enrolled at Beni-Suef University Hospital and randomly assigned to one of four treatment groups (n=100). The primary outcome was the change in intravaginal ejaculatory latency time (IVELT), while secondary outcomes included ejaculatory control and sexual satisfaction, assessed using the Premature Ejaculation Profile Questionnaire (PEPQ). Side effects were also evaluated using multivariate regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PE according to Premature Ejaculation Profile Questionnaire (PEPQ) and the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-V-TR)[12].
* Persistent or recurrent ejaculation within approximately 1 minute of vaginal penetration (confirmed by stopwatch-measured IELT ≤60 seconds at baseline)
* Inability to delay ejaculation during all or nearly all vaginal penetrations
* Negative personal consequences (distress, frustration, avoidance of sexual intimacy)
* PEPQ score ≥11.

  * Age ≥ 20 years.
  * In a stable, monogamous, heterosexual relationship for at least 3 months.
  * Signed informed consent indicating willingness to participate.

Exclusion Criteria:

* Use of PE medications in the preceding 4 weeks.
* Use of hormonal supplements.
* Patients with erectile dysfunction diagnosed by International Index of Erectile Function.
* History of psychiatric or significant physical disorders (in either patient or partner).
* Use of antidepressants, local anesthetic sprays, intracavernosal injections, or psychotherapy within 4 weeks.
* Alcohol or substance abuse.
* Documented hypotension.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 450 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
● Intravaginal Ejaculatory Latency Time: Minimum Value: 0 seconds Maximum Value: No fixed maximum, but usually recorded up to ~30 minutes in clinical studies Interpretation: Lower IELT values indicate worse outcomes, as they reflect shorter ejaculator | 3 months

SECONDARY OUTCOMES:
● Premature Ejaculation Profile Questionnaire (PEPQ): Each item is scored from 1 to 5, and the total score ranges from 4 to 20. Minimum Value: 4 Maximum Value: 20 Higher scores indicate better outcomes | 3 MONTHS
Adverse events | 3 months
  ● Side effects: Adverse effects were evaluated in terms of occurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdellatif A, Elbatanouny A, Ragheb A, Abdelbary A, Eid A, Lotfy AM, Mahmoud O, Youssef M, Abdallah M. Comparative evaluation of safety and efficacy of dapoxetine, silodosin, and citalopram in the management of premature ejaculation: a randomized clinical trial. BMC Urol. 2025 Dec 1;25(1):298. doi: 10.1186/s12894-025-01973-7. PMID 41327131

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT07113145/Prot_SAP_000.pdf